CLINICAL TRIAL: NCT01146613
Title: A Phase 2, Double Blind, Placebo Controlled Trial to Assess the Efficacy of Varenicline Tartrate for Alcohol Dependence in Very Heavy Drinkers
Brief Title: Varenicline for Alcohol Dependence
Acronym: NCIG 003
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIAAA-DTRR-2010-LITTEN-003
Record Dates: First submitted 2010-06-16; First posted 2010-06-17 (Estimated); Results first posted 2014-08-11 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: Alcoholism
Keywords: Alcohol; Alcohol abuse; Alcoholism; Alcohol Dependence; Varenicline; Drinking
MeSH Terms: conditions — Alcoholism | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Varenicline (Active Comparator): Varenicline Tartrate
  Interventions: Drug: Varenicline
- Sugar Pill (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Varenicline — 0.5mg capsules x 2, 2x a day for 12 weeks
  Other Names: Chantix
  Arms: Varenicline
Drug: Placebo — identical matched placebo x 2, 2xday, 13 weeks
  Arms: Sugar Pill

SUMMARY:
The primary objective of this study is to assess the efficacy of varenicline in reducing the proportion of heavy drinking days during the last 8 weeks of treatment in subjects with alcohol dependence confirmed by Diagnostic and Statistical Manual of Mental Disorders-IV-Text Revision (DSM-IV-TR) criteria and who frequently consume 10 or more drinks per drinking day for men and 8 or more drinks for women (designated as "very heavy" drinkers).

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years of age.
2. Have a current (past 12 months) DSM-IV-TR diagnosis of alcohol dependence.
3. Be seeking treatment for alcohol dependence and desire a reduction or cessation of drinking.
4. Be able to verbalize an understanding of the consent form, able to provide written informed consent, verbalize willingness to complete study procedures, able to understand written and oral instructions in English and able to complete the questionnaires required by the protocol.
5. Agree (if the subject is female and of child bearing potential) to use at least one of the following methods of birth control, unless she is surgically sterile, partner is surgically sterile or she is postmenopausal:

   1. oral contraceptives,
   2. contraceptive sponge,
   3. patch,
   4. double barrier (diaphragm/spermicidal or condom/spermicidal),
   5. intrauterine contraceptive system,
   6. levonorgestrel implant,
   7. medroxyprogesterone acetate contraceptive injection,
   8. complete abstinence from sexual intercourse,
   9. hormonal vaginal contraceptive ring, and/or
6. Be able to take oral medication and be willing to adhere to the medication regimen
7. Complete all assessments required at screening and baseline.
8. Provide evidence of stable residence in the last 2 months prior to randomization, have reasonable transportation arrangements to the study site, and have no plans to move within the next 3 months or unresolved legal problems. Subjects must provide contact information of someone, such as a family member, spouse, or significant other, who may be able to contact the subject in case of a missed clinic appointment.
9. Be willing to discontinue the use of nicotine replacement therapies prior to randomization and refrain from using nicotine replacement therapies during the course of the study.
10. Have a blood alcohol content (BAC) by breathalyzer equal to 0.000 when s/he signed the informed consent document.
11. Be someone who in the opinion of the investigator would be expected to complete the study protocol.
12. Agree to the schedule of visits, verbally acknowledge that s/he will be able to attend each scheduled visit, participate in phone visits and that s/he does not have any already scheduled events or a job that may interfere with study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-02; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raye Z. Litten, PhD, Study Director — National Institute on Alcohol Abuse and Alcoholism (NIAAA); Joanne Fertig, PhD, Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA); Daniel E Falk, PhD, Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (7):
- United States (7):
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Dartmouth Medical School, Bedford, New Hampshire
  - Dartmouth Medical School, Hanover, New Hampshire
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
  - University of Virginia, Richmond, Virginia

REFERENCES:
- [Derived] Falk DE, O'Malley SS, Witkiewitz K, Anton RF, Litten RZ, Slater M, Kranzler HR, Mann KF, Hasin DS, Johnson B, Meulien D, Ryan M, Fertig J; Alcohol Clinical Trials Initiative (ACTIVE) Workgroup. Evaluation of Drinking Risk Levels as Outcomes in Alcohol Pharmacotherapy Trials: A Secondary Analysis of 3 Randomized Clinical Trials. JAMA Psychiatry. 2019 Apr 1;76(4):374-381. doi: 10.1001/jamapsychiatry.2018.3079. PMID 30865232
- [Derived] Falk DE, Castle IJ, Ryan M, Fertig J, Litten RZ. Moderators of Varenicline Treatment Effects in a Double-Blind, Placebo-Controlled Trial for Alcohol Dependence: An Exploratory Analysis. J Addict Med. 2015 Jul-Aug;9(4):296-303. doi: 10.1097/ADM.0000000000000133. PMID 26083958
- [Derived] Litten RZ, Ryan ML, Fertig JB, Falk DE, Johnson B, Dunn KE, Green AI, Pettinati HM, Ciraulo DA, Sarid-Segal O, Kampman K, Brunette MF, Strain EC, Tiouririne NA, Ransom J, Scott C, Stout R; NCIG (National Institute on Alcohol Abuse and Alcoholism Clinical Investigations Group) Study Group. A double-blind, placebo-controlled trial assessing the efficacy of varenicline tartrate for alcohol dependence. J Addict Med. 2013 Jul-Aug;7(4):277-86. doi: 10.1097/ADM.0b013e31829623f4. PMID 23728065

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Varenicline | Sugar Pill
Started | 99 | 101
Completed | 92 | 89
Not Completed | 7 | 12
Not completed — Lost to Follow-up | 3 | 8
Not completed — Lack of Efficacy | 0 | 1
Not completed — Death | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 0 | 3
Not completed — schedule conflict | 1 | 0
Not completed — Outpatient detox | 1 | 0

BASELINE CHARACTERISTICS:
Population: One subject (two records) was excluded from analysis due to his dual study participation at two separate clinical sites. Both instances of participation were in the Varenicline arm and both instances were not considered in the mITT population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | Sugar Pill | Total
Number analyzed (Participants) | 97 | 101 | 198
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (11) | 45 (12.3) | 45.5 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 32 | 58
  Male | 71 | 69 | 140
Region of Enrollment [Number; unit: participants]
  United States | 97 | 101 | 198
Drinks per day [Mean (Standard Deviation); unit: drinks per day] | 14 (9.3) | 12.5 (9) | 13 (9)
Drinks per drinking day [Mean (Standard Deviation); unit: drinks per drinking day] | 15.3 (9.6) | 13.6 (9) | 14.4 (9.3)
Percent days abstinent [Mean (Standard Deviation); unit: percent days abstinent] | 7.7 (12.5) | 7.9 (13.6) | 7.8 (13)
Percent heavy drinking days [Mean (Standard Deviation); unit: percent heavy drinking days] | 88.1 (15.8) | 87.2 (16.4) | 87.7 (16.1)
Penn Alcohol Craving Scale Score [Mean (Standard Deviation); unit: score] — PACS Scale Range (0-30) - A higher value score equals more craving.
  score | 17.7 (6.2) | 16.7 (6.8) | 17.2 (6.5)
Alcohol-related consequences score - ImBIBE [Mean (Standard Deviation); unit: score] — ImBIBe - 15 questions (0-60) - Lower score is better The Impact of Beverage Intake on Behavior (ImBIBe) is a 15-item questionnaire in which the subject responds on a 5-point scale to questions on the consequences of alcohol use. This scale was adapted from the Drinker Inventory of Consequences questionnaire based on FDA recommendations on patient reported outcomes (Miller & Tonigen-1995).
  score | 17.8 (9.8) | 16.3 (9.7) | 17 (9.7)
Age of onset of regular drinking [Mean (Standard Deviation); unit: years] — One question asking at what age regular drinking began.
  years | 18.7 (6.1) | 19.3 (5.5) | 19 (5.8)
Gamma-glutamyl transpeptidase (GGT) [Mean (Standard Deviation); unit: IU/L] | 72.9 (123.5) | 70.1 (103.1) | 71.9 (113.3)

OUTCOME MEASURES:

1. Primary Outcome: Weekly Percentage of Heavy Drinking Days
Description: Protocol: The primary outcome measure examines the hypothesis that varenicline will decrease the weekly proportion of heavy drinking days during Study Weeks 2 through 13 as compared to placebo.
Time Frame: Weeks 2-13*
Measure: Mean (Standard Error); unit: percentage of heavy drinking days
Arm/Group | Varenicline | Sugar Pill
Number analyzed (Participants) | 97 | 101
percentage of heavy drinking days | 37.9 (3.6) | 48.4 (3.52)

ADVERSE EVENTS:
Description: AEs were assessed by virtue of an open ended question and by subject report.
Arm/Group | Varenicline | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 2/97 | 2/101
Other Adverse Events (participants affected / at risk) | 88/97 | 90/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=97) | Sugar Pill (N=101)
Gout (General disorders) | 0 (0) | 1 (1)
Hospitalization for a Heniated Disc (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hospitalization for Back Surgery (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Death From Gunshot Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=97) | Sugar Pill (N=101)
constipation (Gastrointestinal disorders) | 9 | 2
Diarrhoea (Gastrointestinal disorders) | 11 | 10
Nausea (Gastrointestinal disorders) | 36 | 18
Vomiting (Gastrointestinal disorders) | 12 | 10
Chest Pain (General disorders) | 0 | 6
Fatigue (General disorders) | 14 | 11
Irritability (General disorders) | 11 | 5
Nasopharyngitis (Infections and infestations) | 6 | 7
Upper respiratory tract infection (Infections and infestations) | 5 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 7
Back Pain (Musculoskeletal and connective tissue disorders) | 6 | 9
Dizziness (Nervous system disorders) | 11 | 6
Dysgeusia (Nervous system disorders) | 6 | 1
Headache (Nervous system disorders) | 26 | 30
Somnolence (Nervous system disorders) | 6 | 13
Abnormal Dreams (Psychiatric disorders) | 27 | 12
Agitation (Psychiatric disorders) | 12 | 16
Anxiety (Psychiatric disorders) | 9 | 8
Depression (Psychiatric disorders) | 7 | 6
Hostility (Psychiatric disorders) | 6 | 4
Insomnia (Psychiatric disorders) | 15 | 12
Rash (Skin and subcutaneous tissue disorders) | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The NIAAA Project Officer is responsible for overseeing the preparation of the main paper summarizing the main findings of the completed Study (the "Main Paper"). No single site data will be published or otherwise disseminated without first consulting and coordinating any such publication or dissemination with the investigators from all stakeholders. Additional manuscripts published after the publication of the Main Paper may be initiated and primarily authored by NIAAA.